CLINICAL TRIAL: NCT00707421
Title: A Randomized Clinical Trial Comparing Preoperative Topical Non-Steroidal Anti-Inflammatory Drugs or Steroids Compared to Placebo With Regard to Clinical Outcomes Following Trabeculectomy.
Brief Title: Usefulness of Topical Non-Steroidal Anti-Inflammatory Drugs or Steroids Before Trabeculectomy and Clinical Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Funding for Research in Ophthalmology (FRO) (Unknown)
Responsible Party: Ingeborg Stalmans, MD, PhD, University Hospitals Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FRO Pre-op Med Trab
Record Dates: First submitted 2008-06-24; First posted 2008-06-30 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Glaucoma; Trabeculectomy; Fibrosis; Intraocular Pressure
MeSH Terms: conditions — Glaucoma; Fibrosis | interventions — Ketorolac; Fluorometholone; Idoxuridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Placebo Comparator): placebo, artificial tears
  Interventions: Drug: artificial lacrimal tears
- 3 (Active Comparator): corticosteroid , CS
  Interventions: Drug: fluorometholone
- 2 (Active Comparator): non-steroidal anti-inflammatory drug, NSAID
  Interventions: Drug: ketorolac acetate

INTERVENTIONS:
Drug: ketorolac acetate
  Other Names: Aculare, Allergan
  Arms: 2
Drug: fluorometholone
  Other Names: FML, Allergan
  Arms: 3
Drug: artificial lacrimal tears
  Other Names: Liquifilm, Allergan
  Arms: 1

SUMMARY:
Antiglaucoma medication have been shown to induce subclinical conjunctival inflammation in a considerable proportion of glaucoma patients. Today, trabeculectomy still remains the gold standard as surgical treatment of medically uncontrolled glaucoma disease. However, this procedure is associated with variable possible complications, of which subconjunctival fibrosis is the most frequent one. The latter results in a non-functional filtering bleb. As a consequence, either additional interventions such as laser suture lysis, needling, bleb revision or additional IOP-lowering medication is necessary. Previous studies demonstrated a benefit of the use of topical steroids postoperatively in reducing inflammation and subsequent subconjunctival fibrosis. In this perspective, we will prospectively explore the usefulness of topical NSAID or corticosteroid therapy preoperatively as compared to placebo in subjects scheduled for first-time trabeculectomy, without interrupting topical antiglaucoma therapy. This will allow us to determine wether the impact of longterm topical antiglaucoma therapy on subclinical conjunctival inflammation which possibly result in postoperative fibrosis and bleb failure can be reversed by anti-inflammatory medication before filtering surgery.

DETAILED DESCRIPTION:
This prospective double-blind randomized placebo-controlled clinical trial was approved by our institutional review board and adheres to the tenets of the Declaration of Helsinki. Patients who agree for the study had to sign an informed consent.

Eligible subjects will be subsequently allocated into one of three topical study medication groups by a computer-based randomisation programme: the placebo group received artificial lacrimal tears (Liquifilm®), the NSAID group a non-steroidal anti-inflammatory drug (Aculare®, ketorolac), and the CS group a corticosteroid (FML®, fluorometholone). All study medication is made by the same pharmaceutical manufacturer (Allergan™), and contained the preservative benzalkonium chloride. Each subject of the 3 study groups will have to take one drop of their study medication four times daily for one month before filtering surgery in addition to their routine antiglaucoma medication. The trabeculectomy technique will be done according to a modified Moorfields procedure by experienced surgeons (IS, TZ)using a standard fornix-based approach.

Patients will be postoperatively examined on days 1 and 2, at weeks 1, 2, and 4, and at months 3, 6, 12, 18 and 24 following trabeculectomy. IOP will be measured by Goldmann applanation tonometry. IOP outcomes will be the observed IOP values and relative (percentage reduction) IOP reduction as compared to baseline at the different postoperative time points. In addition, complete (without additional postoperative medication) and qualified (with and without additional postoperative medication), and number of postoperative additional treatments (needling, laser suture lysis, needling revision) in the study eye will be assessed.

Statistical Analysis

Before the onset of the study, sample size and power calculations are performed. In addition, a randomization programme was set up. A multivariate regression model was used to compare the IOP evolution between the three groups .

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients planned for first-time trabeculectomy willing to comply with the study requirements and having signed informed consent.
* Study subjects have to be diagnosed with glaucoma disease and on maximal medical antiglaucoma medication for at least half a year.

Exclusion Criteria:

* monophthalmic patients
* secondary (e.g. inflammatory) glaucoma
* intake of steroids
* history of recurrent corneal herpes infection (considered as contra-indication for steroids)
* allergy to steroids, NSAID's, or the preservative benzalkonium chloride
* history of previous filtering surgery or any other intraocular surgery except cataract removal
* patients not fulfilling study requirements
* not taking their study group medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of additional IOP-lowering procedures or postoperative medication; Intraocular pressure evolution

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium